CLINICAL TRIAL: NCT01580371
Title: Phase I Clinical Trial to Assess the Safety and Pharmacokinetic Profile of CKD-581 in Patients With Lymphoma or Multiple Myeloma Failed to Standard Therapy
Brief Title: Safety and Pharmacokinetic Profile of CKD-581
Acronym: CKD-581
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 133HL/NHL11L
Record Dates: First submitted 2012-04-16; First posted 2012-04-19 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Lymphoma; Multiple Myeloma
MeSH Terms: conditions — Lymphoma; Multiple Myeloma | interventions — CKD-581; Histone Deacetylase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): CKD-581
  Interventions: Drug: CKD-581

INTERVENTIONS:
Drug: CKD-581 — CKD-581 qd for Day 1, 8 and 15 every 28days/Cycle
  Other Names: Histone Deacetylase Inhibitor

SUMMARY:
This study is to determine the maximum tolerated dose (MTD), dose limiting toxicity (DLT), safety and pharmacokinetics (PK) profile of a single agent CKD-581 injection in patients with Lymphoma failed to standard therapy. The usefulness of the this regimen is evaluated by response rate, progression free survival.

DETAILED DESCRIPTION:
Recently, the role of transcriptional repression through epigenetic modulation in carcinogenesis has been clinically validated with several inhibitors of histone deacetylases and DNA methyltransferases. It has long been recognized that epigenetic alterations of tumor suppressor genes was one of the contributing factors in carcinogenesis. Inhibitors of histone deacetylase (HDAC) de-repress genes that subsequently result in growth inhibition, differentiation and apoptosis of cancer cells. CKD-581 is developed for HDAC inhibitors. Such as to determine the maximum tolerated dose (MTD), dose limiting toxicity (DLT), safety and pharmacokinetics (PK) profile of a single agent CKD-581 injection in patients with Lymphoma failed to standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* 20 years and older
* Histologically or cytologically confirmed Lymphoma or Multiple myeloma that have failed to standard therapy or for which no life prolonging treatment exists
* ECOG(Eastern cooperative oncology) performance status ≤ 2
* Life expectancy 12 weeks
* Hematopoietic: ANC(Absolute Neutrophil Count) ≥ 1,500/mm3, Platelet count(PLT) ≥ 100,000/mm3, Hemoglobin ≥ 9.0g/dL
* Hepatic: Total bilirubin > 1.5×upper limit of normal(except Gilbert's syndrome patients), aspartate aminotransferase(AST) > 3×upper limit of normal, alanine aminotransferase(ALT) > 3×upper limit of normal(AST, ALT ≤ 5.0×ULN in case of liver metastases)
* Renal: serum creatinine ≤ 1.5×upper limit of normal
* Serum calcium ≤ upper limit of normal (If the Multiple myeloma only)
* Signed a written informed consent

Exclusion Criteria:

* Have symptoms with Brain metastases
* History of Ischemic heart disease(e.g., myocardial infarction, unstable angina pectoris) or Clinically significant heart disease such as NYHA Class III and IV Congestive atrial arrhythmias, within 6 months prior to first dose of study drug
* Acute infection or blooding tendencies that would preclude study compliance
* Other psychiatric disorders or other conditions that would preclude study compliance
* Receiving antitumor therapy(surgery, immunotherapy or chemotherapy) within 4 weeks prior to first dose of study drug(6 weeks for nitrosoureas and mitomycin C, 2 weeks for radiation therapy)
* Other concurrent antitumor therapy
* Have Cardiac disease by nature
* Administration history of Histone Deacetylase Inhibitor
* History of Serious hypersensitivity or allergy
* Pregnant or nursing, active serum pregnancy test. Fertile patients must use effective contraception
* Participation in a clinical trial within 4 weeks of first dose of study drug

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-05; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | Up to 28 days (For 1st cycle)

SECONDARY OUTCOMES:
Dose Limiting Toxicity | Up to 28 days (For 1st cycle)
Pharmacokinetics | 0, 0.25, 1, 1.5, 2, 2.25, 2.5, 3, 3.5, 4, 6, 8, 12, 24 hrs post dose(1st cycle Day1, 15)
  PK parameters(AUC, Cmax) of CKD-581 & metabolites
Objective response rate | every 56 days (every 2 cycle)
Progression Free survival | up to progression

CONTACTS AND LOCATIONS:
Overall Officials: Dok Hyun Yoon, Ph.D, Study Chair — 88,Olympic-ro 43-gil, Songpa-gu, Seoul 138-736, Korea
Locations (1):
- ASAN Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No